CLINICAL TRIAL: NCT02919150
Title: Myotonometric Measurement of Myofascial Trigger Points: Reliability, Validity and Sensitivity
Status: Completed | Type: Observational
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: Hospital Nacional de Parapléjicos de Toledo (Other); Universidad San Jorge (Other)
Responsible Party: Sponsor
Other Study IDs: 134a
Record Dates: First submitted 2016-09-27; First posted 2016-09-29 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2016-11

CONDITIONS: Muscle Tone Abnormalities
Keywords: Myofascial Trigger Points; Myotonometry; Isokinetic Dynamometry; Assessment; Reliability

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Myotonometric and isokinetic measurement: Myotonometric assessment: into the site of the latent medial myofascial trigger point of the soleus muscle and distal to the lateral medial myofascial trigger point of the soleus muscle but into the same taut band.
  Isokinetic assessment: triceps surae muscle tone will be quantified by measuring the passive range of motion for ankle dorsiflexion and the resistance to passive ankle dorsiflexion at slow and fast velocity.

SUMMARY:
The aims of this study are:

* To examine the inter-rater reliability to assess myofascial trigger points using a myotonometer
* To determinate the strength of the correlation between myotonometric parameters and isokinetic parameters
* To evaluate the sensitivity of myotonometric measurements to detect the location of myofascial trigger points

DETAILED DESCRIPTION:
Previous researches have used complicated and expensive methods to measure mechanical properties of muscle tone like isokinetic dynamometer.

The purpose of this investigation is to establish the reliability, validity and sensitivity of a myotonometer to assess myofascial trigger points. The results of this study will verify the inter-reliability of a myotonometer device in order to evaluate muscle tone, examine correlations and associations between myotonometric measurements and isokinetic measurements and provide a measurable understanding of the location of myofascial trigger points.

Assessment:

Myoton device is a simple and portable tool to obtain quantitative and objective assessments of mechanical properties of muscle tone.

Isokinetic dynamometric technique is considered a valid biomechanics method to measure muscle tone in non-injured subjects but isokinetic machine is a heavy and expensive equipment.

Outcome measures:

Myotonometric measures will include muscle frequency, decrement (elasticity) and stiffness.

Isokinetic measures will include passive resistive torque to ankle dorsiflexion and dorsiflexion passive range of motion (PROM)

All outcome measures will be evaluated once.

ELIGIBILITY:
Inclusion Criteria:

* Age range 18-55 years.
* Healthy volunteers.
* Presence of a latent medial MTrP of the soleus muscle.
* Being able to provide written informed consent.
* Being able to follow instructions and realize clinical tests.

Exclusion Criteria:

* Any history of ipsilateral lower limb severe injury or intervention (e.g. fracture, surgical intervention).
* Pain or musculoskeletal injury, ligament injury, tendonitis or plantar fasciitis in the ipsilateral leg for six months previous to the evaluation.
* Peripheral or central nervous system neurological disease.
* Altered sensitivity in the studied area.
* Treatment of a myofascial trigger point in the sural triceps in the six months previous to the evaluation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects must be healthy volunteers and will be recruited from the city of Toledo.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Inter-rater reliability of myotonometric measurement | Day 1
  In order to study the interrater reliability of the myoton, two different evaluators assess the muscle tone within two marked points using the myotonometer
Correlation between myotonometric measurement and isokinetic measurement | Day 1
  Relationships among myotonometric parameters and isokinetic parameters
Sensitivity of distinguishing the localisation of myofascial trigger points within the taut band | Day 1
  Ability to identify and differentiate myofascial trigger points and other points within the taut band using the myotonometer

CONTACTS AND LOCATIONS:
Overall Officials: Julio Gomez Soriano, PhD, Study Director — University of Castilla-La Mancha; Carolina Jiménez Sánchez, MSc, Principal Investigator — Universidad San Jorge

IPD SHARING:
Plan to Share IPD: No